CLINICAL TRIAL: NCT06668792
Title: An Open-Label Clinical Study of the Efficacy and Safety of BCD-248 in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: An Open-Label Clinical Study of the Efficacy and Safety of BCD-248 in Patients With Relapsed/Refractory Multiple Myeloma
Acronym: FLAMMINGO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-248-2
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCD-248 (Experimental)
  Interventions: Drug: BCD-248

INTERVENTIONS:
Drug: BCD-248 — subcutaneously

SUMMARY:
The aim of the study is to assess the efficacy and safety of BCD-248 as a therapy for relapsing and/or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Age ≥18 years.
3. Documented diagnosis of multiple myeloma according to the IMWG criteria.
4. Measurable disease at screening.
5. Subjects who received at least 2 lines of therapy for multiple myeloma, including a proteasome inhibitor, an immunomodulatory drug, anti-CD38 therapy.
6. Documented progression according to the IMWG criteria during or after the last line of therapy.
7. Evidence of at least a partial response according to the IMWG criteria to at least 1 previous line of therapy.
8. ECOG score 0-2.

Exclusion Criteria:

1. Subjects who were previously treated with anti-BCMA or anti-CD3 drugs.
2. Use of any investigational medicinal products or medical devices within 30 days or 5 half-lives (whichever is longer) prior to the expected start of the study therapy or planned use of investigational medicinal products or medical devices during participation in this study, except for the use described in this Protocol.
3. Autologous hematopoietic stem cell transplantation within 12 weeks prior to the expected start of the study therapy or a history of allogenic stem cell transplantation, regardless of when it was performed.
4. Planned hematopoietic stem cell transplantation before disease progression during this study.
5. A history of other malignancies within 5 years before screening, excluding squamous and basal cell skin cancers, carcinoma in situ of the cervix or breast, or other malignancies, which, in the opinion of the Investigator, have been adequately treated and have a minimal risk of recurrence within 5 years.
6. Concomitant diseases and/or conditions that significantly increase the risk of AEs during the study:

   * Stable angina pectoris, functional class III-IV.
   * Unstable angina and/or myocardial infarction within less than 6 months before the expected start of the study therapy.
   * Chronic heart failure, NYHA class III-IV;
   * Clinically significant (in the Investigator's opinion) cardiac arrhythmia and conduction disorders that do not respond to the maximum possible antiarrhythmic therapy (therapy should be stable for 4 weeks before the expected start of the study therapy);
   * Moderate to severe asthma, grade III-IV chronic obstructive pulmonary disease, a history of angioedema, severe respiratory failure;
   * Active autoimmune diseases (subjects with type 1 diabetes mellitus and hypothyroidism requiring only hormone replacement therapy, as well as with skin diseases (vitiligo, alopecia, or psoriasis) that do not require systemic therapy are eligible);
   * Any infection within 14 days prior to the expected start of the study therapy, requiring systemic etiotropic therapy or which, in the opinion of the Investigator, may increase the risk of infectious complications;
   * Any other concomitant disease or condition, which, in the Investigator's opinion, significantly increases the risk of AEs in the study.
7. Subjects with amyloidosis.
8. Clinical signs of meningeal involvement of multiple myeloma.
9. HIV infection, active HBV infection, hepatitis C.
10. Major surgery within less than 14 days prior to the expected start of the study therapy, incomplete recovery from surgery, or planned surgery during participation in the study.
11. Pregnancy or breastfeeding, as well as intention to become pregnant or father a child during the study period and within 180 days after receiving the last dose of the IP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate according to IMWG (International Myeloma Working Group) criteria | Up to 24 weeks

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 104 weeks
Complete response (CR) rate according to IMWG criteria | Up to 3.7 years
MRD (minimal residual disease)-negativity rate | Up to 3.7 years
Duration of response | Up to 3.7 years
Time to progression | Up to 3.7 years
Time to response | Up to 3.7 years
Overall survival | Up to 3.7 years
Incidence and characteristics of adverse events | Up to 3.7 years
Cmax after the first administration | up to Day 6
Cmin after the first administration | up to Day 6
AUC0-t after the first administration | up to Day 6
Ctrough | up to 6 months
Soluble BCMA concentration in the blood | Up to 6 months
Proportion of subjects with BAbs | Up to 3 years
Proportion of subjects with NAbs | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (20):
- Russia (20):
  - SBHI of the Kaliningrad region "Central City Clinical Hospital", Kaliningrad
  - SAHI "Republican Clinical Oncology Dispensary of the Ministry of Health of the Republic of Tatarstan named after Professor M.Z. Sigala", Kazan'
  - FSBI of science "Kirov research Institute of Hematology and blood transfusion of the Federal medical and biological Agency", Kirov
  - Regional Government-Owned Publicly Funded Healthcare Institution "Regional Clinical Hospital", Krasnoyarsk
  - Branch of the limited liability company "Hadassah Medical LTD", Moscow
  - City Clinical Hospital №52 of the Department of Health of the City of Moscow, Moscow
  - FSBI "National Medical Research Center of Oncology named after N. N. Blokhin" of the Ministry of Health of the Russian Federation, Moscow
  - JSC "Medsi Group of Companies", Moscow
  - SBI of health care of the city of Moscow city clinical hospital named after S. P. Botkin of the Department of health of the City of Moscow, Moscow
  - State budgetary healthcare Institution of the Moscow Region "Moscow Regional Research Clinical Institute named after M. F. Vladimirsky", Moscow
  - Federal State Budgetary Institution "National Medical Research Center for Radiology" of the Ministry of Health of the Russian Federation, Obninsk
  - SBHI of the Republic of Karelia "Republican Hospital named after V.A. Baranov", Petrozavodsk
  - FSBI "Almazov National Medical Research Centre" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - FSBEI of Higher Education "Samara State Medical University" of the Ministry of Health of the Russian Federation, Samara
  - FSBEI HE "Saratov State Medical University named after V.I. Razumovsky" of the Ministry of Health of Russia, Saratov
  - Private healthcare institution "Clinical hospital "RZD-Medicine" of the city of Smolensk", Smolensk
  - State Budgetary Healthcare Institution "Oncological Dispensary No.2" of the Ministry of Health of the Krasnodar Region, Sochi
  - Public institution "Komi Republican cancer clinic", Syktyvkar
  - FSBEI of Higher Education "Bashkir State Medical University" of the Ministry of Health of the Russian Federation, Ufa
  - State budgetary healthcare institution of the Sverdlovsk region "Sverdlovsk regional clinical hospital №1", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No